CLINICAL TRIAL: NCT06389045
Title: Effect of Propofol Infusion-Based Sedation on Anesthesia-Related Adverse Events in Endoscopic Ultrasonography: A Prospective Observational Study
Brief Title: Propofol Infusion-Based Sedation on Anesthesia-Related Adverse Events in Endoscopic Ultrasonography
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: EUS
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Sedation Complication; Endoscopic Ultrasonography; Procedural Sedation
Keywords: Procedural Sedation; Sedoanalgesia; Endoscopic Ultrosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Procedural Sedation — Profopol Sedation in Endoscopic Ultrasonography

SUMMARY:
Endoscopic ultrasonography (EUS) is an endoscopic procedure performed to investigate conditions affecting the stomach, liver, and bile ducts, as well as for therapeutic interventions. The complexity of EUS can vary significantly, with increased complexity affecting procedure duration, technical success, and the occurrence of adverse events. For the comfort of patients and the success of the procedure, these interventions are typically performed under anesthesia with procedural sedation. To enhance the success rate of the procedure, reduce the risk of side effects, and maximize patient comfort, EUS is generally performed under sedation according to the recommendations of the American Society of Anesthesiologists (ASA). During sedation, the aim is for the patient to be more relaxed and comfortable while maintaining spontaneous respiratory function. Preserving spontaneous respiratory parameters is crucial for procedural safety.

DETAILED DESCRIPTION:
Within the scope of this study, patients undergoing endoscopic ultrasonography (EUS) under anesthesia in the endoscopy unit will be examined. We administered propofol infusion for procedural sedation for patients undergoing therapeutic EUS in our hospital's endoscopy unit. We aimed to evaluate the impact of this sedation method on anesthesia-related adverse events. The primary outcome of this study was to evaluate the anesthesia-related adverse events, which were defined as arrhythmia, hypotension, desaturation, vomiting, undesirable patient movement, coughing, and hiccups during EUS probe insertion. The secondary outcome was defined as the patient's recovery time from anesthesia. In addition, bolus/infusion drug doses used for anesthesia induction and maintenance, demographic data, EUS indications in patients, and comorbidities of patients were recorded.

Vital parameters will be recorded during the procedure and in the recovery unit. Data for the study will be obtained from nurse observation forms and anesthesia records found in patient files. It is an observational study of file scanning nature, which includes information contained in the files.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic ultrasonography (EUS) patients for procedural sedation

Exclusion Criteria:

* Patients who do not sign the consent form.
* Under the age of 18.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo endoscopic ultrasonography (EUS) under procedural sedation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Anesthesia related advers events | during the procedure
  arrhythmia, hypotension, desaturation, vomiting, patient movement, cough during EUS probe insertion, hiccups

SECONDARY OUTCOMES:
recovery time | 1 hour
  Each patient was evaluated using the Post-Anesthetic Discharge Score (PADS)

CONTACTS AND LOCATIONS:
Overall Officials: Caner Genc, M.D., Principal Investigator — Samsun University
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided